CLINICAL TRIAL: NCT02463084
Title: Macronutrient Effects on Alzheimer's Disease: HTN and IR (Hypertension and Insulin Resistance) (MEAL-2)
Brief Title: Macronutrient Effects on Alzheimer's Disease (MEAL-2)
Acronym: MEAL-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 00022512
Record Dates: First submitted 2014-12-19; First posted 2015-06-04 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Prediabetic State; Insulin Resistance; Middle Age; Prehypertension; Mild Cognitive Impairment
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Prehypertension; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Diet (Experimental): Diet intervention consisting of foods with low saturated fats, low glycemic index and low salt
  Interventions: Other: Low Diet
- High Diet (Experimental): Diet intervention consisting of foods with high saturated fats, high glycemic index and high salt
  Interventions: Other: High Diet

INTERVENTIONS:
Other: Low Diet — a 28-day course of 3 meals per day plus 2 snack that are either low in saturated fats, glycemic index and salt.
  Arms: Low Diet
Other: High Diet — a 28-day course of 3 meals per day plus 2 snack that are either high in saturated fats, glycemic index and salt.
  Arms: High Diet

SUMMARY:
This study compares the effects of a one-month diet high in saturated fat (SF), glycemic index (GI), and salt (Na+) to a diet low in these nutritional parameters on memory and other cognitive functions, on MRI measures of brain structure, function, and perfusion, as well as on blood and cerebrospinal fluid levels of amyloid-beta (Aβ), insulin, lipids (total cholesterol, HDL, LDL, oxidized LDL, and triglycerides), cytokines, apolipoprotein E (ApoE), apolipoprotein J, cortisol, soluble low density lipoprotein receptor-related protein (sLRP), and glucose in middle-aged adults (45-65 years of age) with normal cognition or mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be middle-aged (45 to 65 years of age) and will fall on the continuum from healthy (no pre-hypertension or insulin resistance) to pre-hypertensive and insulin resistant (pHAIR).
2. Subjects will not be recruited based on memory status but will have normal memory or memory impairment with a diagnosis of mild cognitive impairment (MCI). Those subjects with MCI will have been assessed by physician and neuropsychologist experts and diagnosed with MCI according to Petersen criteria.

Exclusion Criteria:

1. Diabetes not controlled by diet or exercise; current or previous use of diabetes medications
2. Average systolic blood pressure on three occasions <90 or >139 mm/Hg, diastolic blood pressure <60, or current use of anti-hypertensive medications;
3. Clinically significant elevations in liver function tests as follows: SGOT > 1.5 X ULN, SGPT > 1.5 X ULN, Alkaline Phosphate > 1.5 ULN.
4. Clinically significant elevations in lipid profile as follows: LDL>190, triglycerides>340, or total cholesterol>260 and LDL/HDL ratio >3.0.
5. Significant neurologic disease that might affect cognition, including AD (MCI will be allowed), stroke, Parkinson's disease, multiple sclerosis, or severe head injury with loss of consciousness > 30 minutes or with permanent neurologic sequelae;
6. Significant medical illness or organ failure, such as uncontrolled hypertension or cardiovascular disease, chronic obstructive pulmonary disease, liver disease, or kidney disease;
7. Current use of antipsychotic, anti-depressant, anti-convulsant, anticoagulant, anxiolytic, or sedative medications;
8. Current use of cognition-enhancing medications;
9. Current use of glucocorticoids;
10. Current use of cholesterol-lowering medications, including:

    1. HMG-CoA Reductase Inhibitors [Statins: Atorvastatin (Lipitor), Fluvastatin (Lescol or Lescol EX), Lovastatin, Pravastatin (Pravachol), Rosuvastatin (Crestor), Simvastatin (Zocor)]
    2. Bile Acid Resins [Cholestyramine (Questran), Colestipol, Colesevelam (Welchol)]
    3. Fibric Acids Derivatives [Fenofibrate (Tricor), Gemfibrozil]
    4. Combinations [Amlodipine/Atorvastatin, Niacin/Lovastatin (Advicor), Ezetimibe/Simvastatin (Vytorin)]
    5. Miscellaneous Categories [Ezetimibe (Zetia), Niacin aka Nicotinic acid (Niaspan)
    6. Over-the-counter [Red yeast rice, Niacinamide, Omega 3 fatty acids (fish or flax seed), Slo-Niacin]
11. Common allergies/sensitivities to the following food products: dairy, wheat, gluten, tree nuts or peanuts, eggs, corn, seafood and soy. Other food sensitivities will be assessed on a case-by-case basis.
12. BMI ≤ 18.5
13. Current weight <110 pounds
14. Clinically significant iron deficiency: Hemoglobin <13.5 for white males, <12.2 for white females, <12.5 for black males, and <11.5 for black females.
15. If female, menstruation in the past 12 months or hysterectomy and current hormone replacement therapy medication.
16. Major digestive disorders, absorption issues, or surgeries, including bowel resection, inflammatory bowel diseases (Ulcerative colitis or Crohn's disease), or irritable bowel syndrome (IBS) with a tendency toward diarrhea

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in cerebrospinal fluid levels of Alzheimer's disease biomarkers (CSF beta-amyloid 42) | After 4 week diet intervention
  CSF beta-amyloid 42

SECONDARY OUTCOMES:
Changes in brain structure | After 4 week diet intervention
  MRI entorhinal cortex and white matter volume
Changes in adipose tissue distribution (Change in dual energy x-ray absorptiometry (DEXA) scan and CT measures of central and subcutaneous body fat) | After 4 week diet intervention
  Change in DEXA and CT measures of central and subcutaneous body fat
Changes in cognition (Change in delayed memory and executive function composites) | After 4 week diet intervention
  Change in delayed memory and executive function composites
Change in brain function as measured by MRI | After 4 week diet intervention
  Change in resting state default mode network connectivity
Change in brain perfusion | After 4 week diet intervention
  Change in cerebral perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No